CLINICAL TRIAL: NCT06617325
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Dapirolizumab Pegol in Study Participants With Moderately to Severely Active Systemic Lupus Erythematosus
Brief Title: A Study to Evaluate the Efficacy and Safety of Dapirolizumab Pegol in Study Participants With Moderately to Severely Active Systemic Lupus Erythematosus
Acronym: PHOENYCS FLY
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SL0044; 2019-003407-35 (EudraCT Number); 2023-508191-11 (Registry Identifier: EU Clinical Trials); U1111-1298-3467 (Other: World Health Organization (WHO))
Record Dates: First submitted 2024-09-24; First posted 2024-09-27 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic lupus erythematosus; Dapirolizumab pegol; SLE; DZP
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — dapirolizumab pegol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dapirolizumab pegol (Experimental): Study participants will receive dapriolizumab pegol throughout the Treatment Period.
  Interventions: Drug: DZP
- Placebo (Placebo Comparator): Study participants will receive placebo throughout the Treatment Period.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: DZP — Study participants will receive dapirolizumab pegol (DZP) at prespecified time-points.
  Other Names: CDP7657
  Arms: Dapirolizumab pegol
Other: Placebo — Study participants will receive placebo at prespecified time-points.
  Other Names: PBO
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the ability of dapirolizumab pegol (DZP) as an add-on treatment to standard of care (SOC) medication to achieve clinically relevant long term improvement of moderate to severe disease activity.

ELIGIBILITY:
Inclusion Criteria:

* Study participant must be ≥16 years of age, (≥18 years of age for China), unless restricted by local regulation, at the time of signing the Informed Consent form (ICF)
* Study participants who have moderate to severe disease activity due to either persisting active systemic lupus erythematosus (SLE) or due to an acute worsening of SLE in the scope of frequent relapsing-remitting SLE despite stable standard of care(SOC) medication defined as:

  a. Diagnosed with SLE at least 24 weeks before the Screening Visit by a qualified physician b. Classified by 2019 SLE European League Against Rheumatism/American College of Rheumatology (EULAR/ACR) classification criteria for SLE c. With serological evidence for SLE at Screening as demonstrated by at least 1 of the following: i) Evidence for anti-dsDNA (defined as evidence for anti-dsDNA antibodies in central laboratory) ii) Either complement C3 <lower limit of normal (LLN) OR complement C4 <LLN as measured by central laboratory iii) Antinuclear antibodies with a titer of at least 1:80 confirmed by central laboratory in combination with evidence of at least 1 of the following SLE typical autoantibodies:
  1. Anti-Smith (anti-Sm) antibodies (central laboratory or source verifiable history)
  2. Anti-Sjögren's syndrome antibody A (Anti-SSA) (Ro)/Anti-Sjögren's syndrome antibody B (anti-SSB) (La) autoantibodies (central laboratory)
  3. Historical evidence for anti-dsDNA antibodies
  4. Anti-ribonucleoprotein (RNP) autoantibodies (central laboratory) d. Moderately to severely active defined as:

     * British Isles Lupus Assessment Group Disease Activity Index 2004 (BILAG 2004) Grade B in ≥2 organ systems and/or a BILAG 2004 Grade A in ≥1 organ systems at Screening and Baseline Visit AND
     * Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) ≥6 at the Screening Visit AND
     * SLEDAI-2K without labs ≥4 at Baseline Visit e. Receiving the following standard of care (SOC) medications at stable dose:
     * Antimalarial treatment in combination with glucocorticoids and/or immunosuppressants or as stand-alone treatment if justified OR
     * Treatment with glucocorticoids and/or immunosuppressants if antimalarial treatment is not appropriate (ie, there is documented intolerance in medical history, documented lack of efficacy, contraindications, or lack of availability)

     Exclusion Criteria:
* Study participant has any medical or psychiatric condition (including conditions due to neuropsychiatric SLE) that, in the opinion of the Investigator, could jeopardize or would compromise the study participant's ability to participate in this study. This includes study participants with a life-threatening condition
* Study participant has a history of an anaphylactic reaction to parenteral administration of contrast agents, human or murine proteins, or monoclonal antibodies. This includes systemic reactions due to latex allergy
* Study participant has a history of malignancy, except the following treated cancers: cervical carcinoma in situ (after complete resection [eg, curettage, electrodesiccation] not later than 4 weeks prior to the Screening Visit [V1]), basal cell carcinoma, or dermatological squamous cell carcinoma
* Study participant has a mixed connective tissue disease, scleroderma, and/or overlap syndrome of these diseases with SLE
* Study participant has evidence of human immunodeficiency virus (HIV) infection, agammaglobulinemias, T-cell deficiencies, or human T-cell lymphotropic virus-1 infection at any time prior to or during the study
* Study participant has clinically significant active or latent infection
* Study participant had a reactivated latent infection (eg, cytomegalovirus, herpes simplex virus, or herpes zoster infection) or opportunistic infection (including but not limited to, pneumocystis, cytomegalovirus, or severe herpes zoster infection) within 12 weeks prior to the first study medication infusion (Visit 2) or is currently receiving suppressive therapy for an opportunistic infection
* Study participants who have received live/live attenuated vaccines within 6 weeks prior to the first study medication infusion
* Study participant has used the prohibited medications within the time frame (Wash-Out Period) listed in the Protocol
* Study participant has previously been randomized within this study or has previously been assigned to treatment with dapirolizumab pegol (DZP) in a study evaluating DZP
* Study participant has participated in another study of an investigational medicinal product (IMP) within the previous 12 weeks or 5 half-lives of the IMP whatever is longer, or is currently participating in another study of an IMP
* Study participant has chronic kidney failure stage 4, manifested by estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m2, or serum creatinine >2.5 mg/dL, or participant has proteinuria >3g/day, or protein:creatinine ratio >340 mg/mmol at the Screening Visit

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Achievement of British Isles Lupus Assessment Group Disease Activity Index 2004 (BILAG 2004)-based Composite Lupus Assessment (BICLA) response at Week 48 | Week 48
  A study participant is a BICLA responder if all of the following is fulfilled: a. BILAG 2004 improvement without worsening, defined as BILAG 2004 Grade As at Baseline improved to B/C/D, BILAG 2004 Grade Bs at Baseline improved to C/D, and no BILAG 2004 worsening in other BILAG 2004 organ systems (that had BILAG 2004 Grade C/D/E at Baseline) such that there are no new BILAG 2004 Grades A nor greater than 1 new BILAG 2004 Grade(s) B; and b. No worsening in the Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI- 2K) total score compared to Baseline (defined as no increase in SLEDAI-2K total score); and c. No worsening in the Physician's Global Assessment of Disease (PGA) compared to Baseline defined as ≤10 mm increase on a 100 mm visual analog scale Escape treatment intervention as indicated by investigator until the assessment time point will be defined as an intercurrent event for the primary endpoint leading to non-response from the day after the event onward.

SECONDARY OUTCOMES:
Achievement of SRI 4 response at Week 48 | Week 48
  The Systemic Lupus Erythematosus Responder Index-4 (SRI 4) define responders as (ie, all criteria must be met):
  * Reduction in SLEDAI-2K score of ≥4
  * No shift from BILAG 2004 Grade B, C, D, or E to A post-Baseline
  * No more than 1 shift from BILAG 2004 Grade C, D, or E to B post-Baseline
  * No worsening in the PGA compared to Baseline score; "no worsening" is defined as either no worsening or worsening <10% of the full 100 mm visual analog scale (VAS).
Achievement of prevention of severe BILAG flares (severe BILAG flare-free) through Week 48 | Week 48
  Severe BILAG flare is defined as a BILAG 2004 Grade A in any system due to individual items that are new or worse qualifying for the Grade A.
  Determination of items that are new or worse qualifying for the Grade A will be according to the supplementary information for the numerical scoring of the BILAG-2004 index.
Achievement of LLDAS at Week 40 and maintaining LLDAS at Weeks 44 and 48 | Week 40 to Week 48
  Low lupus disease activity state (LLDAS) is defined as:
  * No significant disease activity as per Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K); SLEDAI-2K score ≤4 with no activity in major organ systems (renal, central nervous system (CNS), cardiopulmonary, vasculitis, fever)
  * No new and/or worsening disease activity defined as no SLEDAI-2K component documented as present that was not documented present at previous visit
  * Physician's Global Assessment of Disease (PGA) ≤33 mm
  * Prednisone equivalent systemic dose for systemic lupus erythematosus (SLE) indication ≤7.5 mg per day
  * Stable standard maintenance doses of immunosuppressive drugs as allowed by protocol
Change from Baseline to Week 48 in the FATIGUE-PRO Total score | From Baseline to Week 48
  The FATIGUE-PRO (Fatigue patient-reported outcome) is a PRO instrument measuring fatigue, a core symptom of SLE, developed using qualitative and quantitative research conducted in patients with SLE. It is composed of 31 items covering 3 domains: Physical Fatigue (items 1-9), Mental and Cognitive Fatigue (items 10-20), and Susceptibility to Fatigue (items 21-31). The study participant is asked to score each fatigue item based on how frequently they experienced the item during the past 7 days using the following response options: 1=none of the time; 2=a little of the time; 3=some of the time; 4=most of the time; 5=all of the time.
Percentage of participants having a reduction in glucocorticoid dose from >7.5mg/day prednisone-equivalent dose at Baseline to ≤7.5mg/day at Week 36 and maintained through Week 48 | From Baseline to Week 48
  The achievement of a reduction in glucocorticoid dose from >7.5mg/day prednisone equivalent dose at Baseline to ≤7.5mg/day prednisone equivalent at Week 36 and maintained through Week 48 will be assessed.
Achievement of BILAG 2004 improvement without worsening at Week 48 | Week 48
  BILAG 2004 improvement without worsening can be defined as A scores at Baseline improved to B, C or D; B scores improved to C or D; no new A scores and ≤1 new B.
Change from Baseline in PGA at Week 48 | From Baseline to Week 48
  Physician's Global Assessment of Disease (PGA), the investigator will rate the overall status of the study participant. The PGA of disease activity used will be a 100 mm linear scale without anchors. The very far left end is 'very good, asymptomatic and no limitation of normal activities'; the very far right end indicates 'severe disease'.
Achievement of prevention of moderate/severe BILAG flares (moderate/severe BILAG flare-free) through Week 48 | During Treatment Period up to Week 48
  A BILAG severe flare is defined as a BILAG 2004 Grade A in any system due to individual items that are new or worse qualifying for the Grade A. Determination of items that are new or worse qualifying for the Grade A will be according to the supplementary information for the numerical scoring of the BILAG-2004 index.
  A BILAG moderate flare is defined as 2 or more BILAG 2004 Grade Bs due to individual items that are new or worse since previous visit and are qualifying for the Grade B in any system. Determination of items that are new or worse qualifying for the Grade B will be according to the supplementary information for the numerical scoring of the BILAG-2004 index.
Change from Baseline in SLEDAI-2K at Week 48 | From Baseline to Week 48
  SLEDAI-2K measures disease activity. Disease activity in the 30 days prior to and at the time point of the assessment shall be considered. It is a global index and includes 24 clinical symptoms and laboratory variables that are weighted by the type of manifestation, but not by severity or dynamic of the individual item. The total score falls between 0 and 105, with higher scores representing increased disease activity.
Change from Baseline in FACIT-Fatigue score at Week 48 | From Baseline to Week 48
  The FACIT (Functional Assessment of Chronic Illness Therapy)-Fatigue scale is a patient-reported outcome (PRO) measure assessing symptoms and impacts of fatigue originally developed in patients with cancer (Cella et al, 2002). It is composed of 13 items, all scored from 0 (Not at all) to 4 (Very much), and uses a recall period of the past 7 days. The FACIT-Fatigue score ranges from 0 to 52 with 0 being the worst possible score and 52 being the best possible score (lowest level of fatigue). To obtain a score from 0 to 52, all negatively worded questions have to be recoded, so that responses range from worst (0) to the best (4) outcome.
Percentage of participants with treatment-emergent adverse events (TEAEs) during the study | From Baseline until Safety Follow-Up (up to Week 54)
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study medication, whether or not considered related to the study medication.
Percentage of participants with serious treatment-emergent adverse events during the study | From Baseline until Safety Follow-Up (up to Week 54)
  A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose:
  1. Results in death
  2. Is life-threatening
  3. Requires inpatient hospitalization or prolongation of existing hospitalization
  4. Results in persistent disability/incapacity
  5. Is a congenital anomaly/birth defect
  6. Is an Important medical event
Percentage of participants with treatment-emergent adverse events of special interest during the study | From Baseline until Safety Follow-Up (up to Week 54)
  An adverse event of special interest is any adverse event (AE) that a regulatory authority has mandated be reported on an expedited basis, regardless of the seriousness, expectedness, or relatedness of the AE to the administration of a UCB product/compound.
Percentage of participants with treatment-emergent adverse events of special monitoring during the study | From Baseline until Safety Follow-Up (up to Week 54)
  An adverse event of special monitoring is a product-specific adverse event (AE), adverse reaction, or safety topic considered as requiring special monitoring by UCB.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (202):
- United States (55):
  - Sl0044 50058, Avondale, Arizona
  - Sl0044 50550, Chandler, Arizona
  - Sl0044 50713, Gilbert, Arizona
  - Sl0044 50662, Glendale, Arizona
  - Sl0044 50052, Phoenix, Arizona
  - Sl0044 50670, Searcy, Arkansas
  - Sl0044 50257, La Jolla, California
  - Sl0044 50275, La Palma, California
  - Sl0044 50755, Los Alamitos, California
  - Sl0044 50258, Los Angeles, California
  - Sl0044 50725, Menifee, California
  - Sl0044 50340, Orange, California
  - Sl0044 50316, San Leandro, California
  - Sl0044 50719, Aurora, Colorado
  - Sl0044 50239, Brandon, Florida
  - Sl0044 50630, Clearwater, Florida
  - Sl0044 50747, Coral Gables, Florida
  - Sl0044 50751, Coral Gables, Florida
  - Sl0044 50362, Gainesville, Florida
  - Sl0044 50763, Margate, Florida
  - Sl0044 50735, Miami, Florida
  - Sl0044 50681, Miami, Florida
  - Sl0044 50324, Plantation, Florida
  - Sl0044 50698, Tampa, Florida
  - Sl0044 50585, Winter Park, Florida
  - Sl0044 50566, Gainesville, Georgia
  - Sl0044 50659, Marietta, Georgia
  - Sl0044 50699, Chicago, Illinois
  - Sl0044 50717, Willowbrook, Illinois
  - Sl0044 50748, New Albany, Indiana
  - Sl0044 50074, Kansas City, Kansas
  - Sl0044 50586, Louisville, Kentucky
  - Sl0044 50023, Baton Rouge, Louisiana
  - Sl0044 50285, Lake Charles, Louisiana
  - Sl0044 50660, New Orleans, Louisiana
  - Sl0044 50730, Rockville, Maryland
  - Sl0044 50219, Detroit, Michigan
  - Sl0044 50682, Kansas City, Missouri
  - Sl0044 50010, Brooklyn, New York
  - Sl0044 50264, Manhasset, New York
  - Sl0044 50077, New York, New York
  - Sl0044 50241, Syracuse, New York
  - Sl0044 50238, Charlotte, North Carolina
  - Sl0044 50365, Pittsburgh, Pennsylvania
  - Sl0044 50001, Jackson, Tennessee
  - Sl0044 50693, Murfreesboro, Tennessee
  - Sl0044 50562, Allen, Texas
  - Sl0044 50738, Bellaire, Texas
  - Sl0044 50673, Fort Worth, Texas
  - Sl0044 50723, Houston, Texas
  - Sl0044 50688, Houston, Texas
  - Sl0044 50696, Houston, Texas
  - Sl0044 50718, Mansfield, Texas
  - Sl0044 50036, Mesquite, Texas
  - Sl0044 50061, Spokane Valley, Washington
- Argentina (7):
  - Sl0044 60004, C.a.b.a
  - Sl0044 60002, Capital Federal
  - Sl0044 60024, Córdoba
  - Sl0044 60029, Mendoza
  - Sl0044 60003, Quilmes
  - Sl0044 60011, San Juan
  - Sl0044 60014, San Miguel de Tucumán
- Belgium (2):
  - Sl0044 40002, Leuven
  - Sl0044 40060, Liège
- Canada (2):
  - Sl0044 50259, Rimouski
  - Sl0044 50045, Toronto
- Sl0044 60018, Santiago, Chile
- China (36):
  - Sl0044 20293, Baotou
  - Sl0044 20128, Beijing
  - Sl0044 20157, Beijing
  - Sl0044 20173, Beijing
  - Sl0044 20201, Bengbu
  - Sl0044 20291, Changchun
  - Sl0044 20342, Changchun
  - Sl0044 20295, Changsha
  - Sl0044 20186, Changzhou
  - Sl0044 20137, Chengdu
  - Sl0044 20019, Guangzhou
  - Sl0044 20360, Guangzhou
  - Sl0044 20290, Guilin
  - Sl0044 20271, Haikou
  - Sl0044 20296, Hangzhou
  - Sl0044 20185, Jinan
  - Sl0044 20364, Jiujiang
  - Sl0044 20192, Nanchang
  - Sl0044 20024, Nanjing
  - Sl0044 20331, Nanning
  - Sl0044 20272, Pingxiang
  - Sl0044 20020, Shanghai
  - Sl0044 20172, Shanghai
  - Sl0044 20346, Shantou
  - Sl0044 20363, Shijiazhuang
  - Sl0044 20204, Suzhou
  - Sl0044 20136, Tianjin
  - Sl0044 20275, Urumuqi
  - Sl0044 20025, Wenzhou
  - Sl0044 20180, Wuhan
  - Sl0044 20270, Wuhan
  - Sl0044 20274, Xi'an
  - Sl0044 20341, Xiamen
  - Sl0044 20273, Yangzhou
  - Sl0044 20132, Zhengzhou
  - Sl0044 20361, Zhuzhou
- Denmark (2):
  - Sl0044 40513, Copenhagen
  - Sl0044 40489, Odense
- France (2):
  - Sl0044 40848, Le Mans
  - Sl0044 40506, Montpellier
- Germany (13):
  - Sl0044 40386, Cologne
  - Sl0044 40716, Cologne
  - Sl0044 40322, Dessau
  - Sl0044 40356, Dresden
  - Sl0044 40072, Freiburg im Breisgau
  - Sl0044 40717, Greifswald
  - Sl0044 40027, Herne
  - Sl0044 40139, Jena
  - Sl0044 40078, Leipzig
  - Sl0044 40854, Mainz
  - Sl0044 40815, München
  - Sl0044 40402, Tübingen
  - Sl0044 40715, Vogelsang-gommern
- Greece (4):
  - Sl0044 40376, Athens
  - Sl0044 40501, Athens
  - Sl0044 40377, Heraklion
  - Sl0044 40507, Larissa
- Italy (9):
  - Sl0044 40816, Brescia
  - Sl0044 40514, Genova
  - Sl0044 40291, Milan
  - Sl0044 40471, Milan
  - Sl0044 40509, Padua
  - Sl0044 40176, Pisa
  - Sl0044 40148, Roma
  - Sl0044 40675, Roma
  - Sl0044 40830, Rozzano
- Japan (24):
  - Sl0044 20035, Bunkyō City
  - Sl0044 20196, Bunkyō City
  - Sl0044 20279, Bunkyō City
  - Sl0044 20030, Chūōku
  - Sl0044 20281, Fukuoka
  - Sl0044 20039, Kawagoe
  - Sl0044 20045, Kita-gun
  - Sl0044 20065, Kitakyushu
  - Sl0044 20301, Kurashiki
  - Sl0044 20069, Meguro-ku
  - Sl0044 20071, Nagasaki
  - Sl0044 20287, Nagoya
  - Sl0044 20084, Saga
  - Sl0044 20283, Sagamihara
  - Sl0044 20031, Sapporo
  - Sl0044 20042, Sasebo
  - Sl0044 20171, Sendai
  - Sl0044 20076, Shinjuku-ku
  - Sl0044 20285, Shinjuku-ku
  - Sl0044 20288, Shinjuku-ku
  - Sl0044 20277, Suita
  - Sl0044 20032, Suita-shi
  - Sl0044 20278, Tsu
  - Sl0044 20276, Yoshida-gun
- Netherlands (3):
  - Sl0044 40838, Amsterdam
  - Sl0044 40292, Groningen
  - Sl0044 40565, Maastricht
- Peru (2):
  - Sl0044 60026, Arequipa
  - Sl0044 60009, Surco
- Poland (10):
  - Sl0044 40398, Katowice
  - Sl0044 40795, Katowice
  - Sl0044 40502, Krakow
  - Sl0044 40037, Lublin
  - Sl0044 40044, Poznan
  - Sl0044 40821, Poznan
  - Sl0044 40097, Warsaw
  - Sl0044 40098, Warsaw
  - Sl0044 40397, Wroclaw
  - Sl0044 40481, Wroclaw
- Puerto Rico (2):
  - Sl0044 50671, Caguas
  - Sl0044 50683, San Juan
- Serbia (4):
  - Sl0044 40730, Belgrade
  - Sl0044 40466, Kragujevac
  - Sl0044 40861, Niška Banja
  - Sl0044 40392, Novi Sad
- South Korea (3):
  - Sl0044 20141, Busan
  - Sl0044 20104, Seoul
  - Sl0044 20092, Suwon
- Spain (13):
  - Sl0044 40045, A Coruña
  - Sl0044 40826, Badajoz
  - Sl0044 40159, Barcelona
  - Sl0044 40160, Barcelona
  - Sl0044 40839, Castellon
  - Sl0044 40857, Madrid
  - Sl0044 40341, Málaga
  - Sl0044 40521, Mérida
  - Sl0044 40101, Sabadell
  - Sl0044 40853, Santiago de Compostela
  - Sl0044 40049, Seville
  - Sl0044 40103, Seville
  - Sl0044 40106, Seville
- Taiwan (6):
  - Sl0044 20330, New Taipei City
  - Sl0044 20080, Taichung
  - Sl0044 20142, Taichung
  - Sl0044 20086, Taipei
  - Sl0044 20099, Taipei
  - Sl0044 20082, Taoyuan
- United Kingdom (2):
  - Sl0044 40847, Bath
  - Sl0044 40281, Leeds

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://www.Vivli.org